CLINICAL TRIAL: NCT01205334
Title: Phase I/II Administration of CMV (Cytomegalovirus)-Specific Cytotoxic T Cells in Patients With Glioblastoma Multiforme (COGLI)
Brief Title: Administration of CMV-Specific Cytotoxic T Cells in Patients With Glioblastoma Multiforme
Acronym: COGLI
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: poor accrual
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other); The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Nabil Ahmed, Assistant Professor Pediatric Hematology/Oncology Center for Cell and Gene Therapy, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 26901-COGLI
Record Dates: First submitted 2010-09-17; First posted 2010-09-20 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2013-08

CONDITIONS: Glioblastoma Multiforme; GBM; Brain Cancer
Keywords: Glioblastoma multiforme; GBM; Brain Cancer; CTL
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Autologous CMV-specific CTL (Experimental): The patient will receive one of the following doses:
  * 1.5x10^7 cells/m2
  * 4.5x10^7 cells/m2
  * 1.5x10^8 cells/m2
  Interventions: Biological: Autologous CMV-specific CTL

INTERVENTIONS:
Biological: Autologous CMV-specific CTL — CMV-specific T cells will be given by intravenous injection over 1-10 minutes through either a peripheral or a central line with a minimum 20g cannula. The expected volume will be 1-50 cc.
  At the discretion of the attending physician, subjects can receive repeat infusions of modified T cells at the same dose level as long as they do not have progressive disease (up to a maximum of 6 doses and the minimum interval between repeat infusions is 6 weeks). Infusion procedures and follow-up will be identical to those for the first infusion. Patients, who receive additional doses of CTLs will be monitored exactly like after the 1st CTL infusion.
  Other Names: Cytomegalovirus-specific cytotoxic T-Lymphocytes

SUMMARY:
Patients have a type of brain cancer called glioblastoma multiforme. Because most GBMs come back after standard therapy, patients are being asked to volunteer to take part in a research study using special immune cells. They may have already thought about being in this study.

Some patients with GBM show evidence of infection with a virus called Cytomegalovirus before the time of their diagnosis. CMV is found in the cancer cells of some patients with GBM, suggesting that it may play a role in causing the disease. The cancer cells infected by CMV are able to hide from the body's immune system and escape destruction. We want to see if special white blood cells, called T cells, that have been trained to recognize and kill special parts of CMV infected cells can survive in the blood and affect the tumor.

We have used this sort of therapy to treat different types of cancer that are positive for other viruses and have had variable results. Some patients have had responses others did not. It is not possible for us to predict if this treatment will work for GBM.

The purpose of this study is to find the largest safe dose of CMV-T cells, to learn what the side effects are, and to see whether this therapy might help patients with GBM.

DETAILED DESCRIPTION:
To generate CMV-T cells we put a specially produced carrier virus (adenovirus) that carries one CMV gene into the patient's blood monocytes or dendritic cells. These cells are then used to train the patient's T cells to kill cells with CMV on their surface. We then grow these CMV-T cells by more stimulations with Epstein-Barr virus (EBV)infected cells from the patient's blood, which also contain the adenovirus with the CMV gene.

When the patient enrolls on this study, they will be assigned a dose of CMV-T cells.

The patient will be given an injection of cells into the vein through an IV line at the assigned dose. The patient will be followed in the clinic after the injection for 1 to 4 hours.

If after a 6 week evaluation period after the infusion, the patient seems to be experiencing a benefit (tumor regression confirmed by radiological studies, physical exam and/or symptoms), they may be able to receive up to six additional doses of the T cells if they wish. These additional infusions would be at least 1 to 3 months apart and at the same dose level they received the first time.

Medical tests before treatment--

Before being treated, the patient will receive a series of standard medical tests: Physical exam, Pregnancy test (if applicable), Blood tests to measure blood cells, kidney and liver function, Measurements of your tumor by routine imaging studies

Medical tests during and after treatment--

The patient will receive standard medical tests when getting the infusions and after: Physical exams, Blood tests to measure blood cells, kidney and liver function, Measurements of your tumor by routine imaging studies 6 weeks after the infusion

To learn more about the way the CMV-T cells are working and how long they last in the body, blood will be taken on the day of the T-cell infusion, before and at the end of the T-cell infusion, 1, 2, 4 and 6 weeks after the T-cell infusion and every 3 months for 1 year.

Total time participation for this study will be 1 year.

ELIGIBILITY:
INCLUSION CRITERIA:

* Histopathological verification of glioblastoma multiforme (GBM: WHO grade IV) in remission (Group A) or with active disease (Group B).
* CMV-positive GBM
* CMV seropositive
* Life expectancy 6 weeks or greater
* Karnofsky/Lansky score 50 or greater
* Patient or parent/guardian capable of providing informed consent
* Bilirubin less than 1.5x upper limit of normal, AST less than 3x upper limit of normal, serum creatinine less than 1.5x normal and Hgb 8.0 g/dL or greater
* Pulse oximetry of 90% or greater on room air
* Sexually active patients must be willing to utilize one of the more effective birth control methods for 6 months after the CTL infusion. The male partner should use a condom.
* Patients should have been off other investigational antineoplastic therapy for one month prior to entry in this study.
* Informed consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent.

EXCLUSION CRITERIA:

* Severe intercurrent infection
* Known HIV positivity
* Pregnant or lactating
* History of hypersensitivity reactions to murine protein-containing products.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-11; Primary Completion 2012-01 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Number of subjects with dose limiting toxicity | 6 weeks
  The main aim will be to collect information about the maximum tolerated dosage to evaluate the safety of escalating doses of autologous CMV-specific cytotoxic T-lymphocytes (CTL) in patients with CMV-positive Glioblastoma multiforme (GBM)

SECONDARY OUTCOMES:
Patients with a decrease in disease after the CTL infusion | 6 weeks
  To evaluate the effects of CMV-specific CTL on measurable disease.
Area under the growth curves (AUC) over time for T cell frequencies | 1 year
  To measure the survival and function of CMV-specific CTL in vivo.

CONTACTS AND LOCATIONS:
Overall Officials: Nabil M. Ahmed, MD, Principal Investigator — Center for Cell and Gene Therapy, Baylor College of Medicine
Locations (2):
- United States (2):
  - Texas Children's Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas